CLINICAL TRIAL: NCT02918591
Title: The Physiological and Cardiovascular Effects of Empagliflozine in Type 2 Diabetes
Brief Title: Cardiovascular Effects of Empagliflozine
Acronym: EMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Professor, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0049-16 WOMC
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozine (Experimental): All type 2 diabetic participant will be treated during 2 month with Empagliflozine 10 to 25 mg daily during 2 month.
  Interventions: Drug: Empagliflozine

INTERVENTIONS:
Drug: Empagliflozine — All 6type 2 diabetic participant will receive treatment with Empagliflozine during 2 month
  Other Names: EMP

SUMMARY:
It has been shown that in patients with type 2 diabetes (T2D) at high risk for cardiovascular disease (CVD) who received Empagliflozine as compared with placebo had a lower rate of death from cardiovascular causes, non-fatal MI, or non-fatal strokes as well as death from any cause and hospitalization for heart failure.

This lower incidence of cardiovascular disease in individuals treated with selective inhibitor of renal sodium-glucose co-transporters (SGLTs) has been associated with reduction of blood levels of fibroblast growth factor 23 (FGF23) and with increase of blood levels of Klotho.

Therefore we will investigate the blood levels of fibroblast growth factor 23 (FGF23) and of Klotho in type 2 diabetic patients treated with Empagliflozine The investigators anticipate that patients treated with Empagliflozine will have decreased levels of FGF23 and increased levels of Klotho which would provide a good explanation for the beneficial cardiovascular effects of selective inhibitors of renal sodium-glucose co-transporters (SGLTs)

DETAILED DESCRIPTION:
Recently it was shown that in patients with type 2 diabetes at high risk for cardiovascular disease (CVD) who received Empagliflozine as compared with placebo had a lower rate of death from cardiovascular causes, non-fatal MI, or non-fatal strokes as well as death from any cause and hospitalization for heart failure Empagliflozine is a selective inhibitor of renal sodium-glucose co-transporters (SGLTs) that has been approved for treatment of type 2 diabetes. It is associated with weight loss, reduction in blood pressure without an increase in heart rate, and improves markers of arterial stiffness and vascular resistance, visceral adiposity, albuminuria and urate.

Renal sodium-glucose cotransporter (SGLT2) resides in the proximal tubule (PT).The latter is anatomically exposed to the initial glomerular filtrate. Therefore the proximal tubule (PT) cells play a variety of roles amongst which are receptor mediated protein endocytosis, reabsorption of sodium, glucose and phosphate At steady state approximately 85% of the filtered phosphate Pi load is reabsorbed by the kidney through sodium phosphate transporters found in the apical membrane of the proximal tubule cells.

These transporters are also affected by fibroblast growth factor 23 (FGF23). Fibroblast growth factor 23 (FGF23) is a hormone that is mainly secreted by osteocytes and osteoblasts in bone, and the levels of FGF23 increase significantly at the very early stages of chronic kidney disease (CKD) and may play a critical role in mineral ion disorders and bone metabolism in these patients.

Recent publications have also shown that FGF23 and its cofactor, Klotho, may play an independent role in directly regulating bone mineralization instead of producing a systematic effect. It augments phosphaturia by affecting sodium phosphate co transporters: mainly :NaP2a Fibroblast growth factor 23 (FGF23) FGF23 binds to a receptor complex consisting of FGFR1, 3 or 4 and α Klotho and activates ERK1/2 leading to internalization and degradation of NaP2a.

Klotho a transmembrane protein identified as an aging suppressor protein , expressed mainly in the distal tubule and to a lesser extent in the PTC serves as a co-receptor along with FGF receptor in the binding of FGF23 in the DCT It is found mainly in kidney distal tubular epithelium, parathyroid gland, epithelial cells of the choroid plexus in the brain and human vascular tissue .Recently it was demonstrated in the PCT as well.

Higher FGF23 levels were found to be associated with all cause mortality in patients with end stage renal disease, on dialysis, with CKD stages 2-4 and in the general population FGF23 has numerous adverse effects which might contribute to CVD: It is associated with abnormal left ventricular geometry, including higher left ventricular mass, higher left ventricular mass to volume ratio, greater risk of remodeling and of atrial fibrillation in. It also activates the renin angiotensin system and promotes sodium reabsorption in the distal tubule of the kidney contributing to volume overload and hypertension Reduction in Klotho's levels has been observed in normal aging and in renal disease, diabetes mellitus and hypertension .

Klotho also exists in a secreted soluble form and as such has distinct actions. The secreted form increases nitric oxide (NO) availability, and protects against endothelial dysfunction. It possesses ant oxidative action as demonstrated in spontaneous hypertensive rats. Chronic kidney disease mice overexpressing Klotho demonstrate almost no aortic calcification.

The complex Klotho/ FGF23 induces urinary phosphate excretion ,reduces serum levels of 1,25 (OH)Vit D and inhibits secretion of PTH .

Enhanced phosphaturia ameliorates vascular calcification. Indeed vessel produced Klotho is an endogenous inhibitor of calcification.

Recently Dapagliflozine a renal sodium-glucose cotransporter SGLT2 inhibitor has demonstrated an enhanced ERK phosphorylation in cell culture of colon cancer If such phosphorylation occurs in ERK in renal proximal tubule cells than this phosphorylation would increase internalization and degradation of NaP2a leading in turn to hypophosphatemia and a decrease in FGF23 levels and increase of Klotho Therefore the investigators will search the blood levels of fibroblast growth factor 23 (FGF23) and of Klotho in type 2 diabetic patients treated with Empagliflozine

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* HbA1C:7.5-10.
* Age>18 years-80 years
* Cardiovascular risk factor: Ischemic heart disease (IHD)
* Status Post Myocardial Infarct (SPMI),
* Angina Pectoris (AP), stable, unstable AP, Peripheral vascular disease (PVD),
* Cerebro vascular accident (CVA), all > 6 month
* Chronic renal failure (CRF),
* e-GFR > 50 ml/min
* Patients will be required to be on stable glucose-lowering therapy for at least 12 weeks before entering the study.

Exclusion Criteria:

* Age<18 years
* Pregnanacy,breast-feeding.
* eGFR < 45mg/dl
* Type1 Diabetes
* Active urogenital infection , or an infection in the last 6 months.
* Recurrent UTI or genital infections.
* SGLT2 treatment.
* History of ketoacidosis.
* Pulmonary embolism/DVT during the last year.
* Malignancy active, (during the last 10 years).
* Steroid use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of Soluble Klotho | up to 2 months
  The blood levels of soluble Klotho will be quantified at baseline after one month and after two month of treatments with Empagliflozine

SECONDARY OUTCOMES:
Change of Fibroblast growth factor 23 (FGF23) | up to 2 months
  The blood levels of FGF23 will be quantified at baseline after one month and after two month of treatment with Empagliflozine
Change of 1,25 (OH)Vit D | up to 2 months
  The blood levels of 1,25 (OH)Vit D will be quantified at baseline after one month and after two month of treatment with Empagliflozine
Change of Parathyroid Hormone (PTH) | up to 2 months
  The blood levels of PTH will be quantified at baseline after one month and after two month of treatment with Empagliflozine
Change of Glomerular Filtration Rate (eGFR) | up to 2 months
  The levels of eGFR will be quantified at baseline after one month and after two month of treatment with Empagliflozine
Change of Blood Chemistry | up to 2 months
  The blood chemistry will be quantified at baseline after one month and after two month of treatment with Empagliflozine
Change of HbA1c | up to 2 months
  HbA1c will be quantified at baseline after one month and after two month of treatment with Empagliflozine

IPD SHARING:
Plan to Share IPD: No